CLINICAL TRIAL: NCT03499483
Title: A Phase IV Open-label Evaluation of Safety, Tolerability, and Acceptability of a Fixed-dose Formulation of Bictegravir, Emtricitabine/Tenofovir Alafenamide (B/F/TAF) for Non-occupational Prophylaxis Following Potential Exposure to HIV-1
Brief Title: Biktarvy for Non-Occupational Post-Exposure Prophylaxis (nPEP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fenway Community Health (Other)
Responsible Party: Principal Investigator, Kenneth H. Mayer, MD, Medical Research Director, Co-Chair TFI, Fenway Community Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1141260-1
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: HIV Prevention
Keywords: Post-Exposure-Prophylaxis
MeSH Terms: interventions — bictegravir; emtricitabine tenofovir alafenamide

STUDY DESIGN:
Intervention Model Description: Open Label single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open Label Biktarvy (Experimental): Single arm all participants receive open label study product intervention.
  Interventions: Drug: bictegravir

INTERVENTIONS:
Drug: bictegravir — Single One Pill Formulation of bictegravir, emtricitabine/tenofovir alafenamide (Bictarvy) to be taken once daily orally for a period of 28 days.
  Other Names: emtricitabine/tenofovir alafenamide

SUMMARY:
Study will evaluate the safety and tolerability of once daily Biktarvy for 28 days for prevention of HIV infection in HIV-1-seronegative adults after high-risk sexual contact. (non-occupational post exposure prophylaxis - nPEP)

DETAILED DESCRIPTION:
Non-randomized, open label single arm trial conducted at Fenway Health as a single site. 100 subjects will be enrolled following a high risk sexual exposure in which HIV exposure is a concern. Each person will be provided with detailed informed consent and if they agree, will receive a 28 day regimen of BIC/F/TAF (Biktary) in a single fixed-dose tablet. Subjects will be seen for 3 visits over a period of four months in which assessments will be done to evaluate safety of product, tolerability of product and HIV status. All subjects will be compared to historical controls in the previous one daily TDF-based nPEP studies which were conducted at Fenway Health.

ELIGIBILITY:
Inclusion Criteria:

1. > Age of 18 at time of first visit.
2. HIV uninfected
3. Willing and able to provide written informed consent.
4. Willing and able to provide adequate locator information.
5. Willing and able to return to all study visits.
6. Willing to participate in all study procedures.
7. Childbearing age: Willing to use contraception for as long as they are on study medication plus 7 days after. (Appendix A: list of approved contraception).
8. Possible sexual exposure to HIV-1, recent enough to permit receiving the first dose of study medication within 72 hours from the end of the exposure. A possible exposure could include:

   1. Condomless anal, vaginal, oral, or mucosal (e.g. conjunctival) exposure to ejaculate from a partner who is HIV-1 infected or high risk for HIV infection and of unknown HIV-1 serostatus (may include protected sexual exposure with condom failure, breakage or slippage); or
   2. Condomless penile exposure to cervicovaginal secretions or anorectal secretions from a partner who is HIV-1 infected or high risk for HIV infection and of unknown HIV-1 serostatus (may include protected sexual exposure with condom failure, breakage or slippage)

Exclusion Criteria:

1. An active psychiatric illness or active drug or alcohol abuse that, in the opinion of the investigator, could prevent compliance with study procedures.
2. Pregnancy and/or breastfeeding.
3. People who are actively trying to become pregnant.
4. Acute or chronic hepatitis B infection.
5. Acute or chronic renal disease.
6. Creatinine clearance at or below 30 mL/min (Cockcroft-Gault0 Known intolerance or allergy to tenofovir disoproxil fumarate, tenofovir alafenamide, emtricitabine, or bictegravir.

8. Currently taking or plans to take prohibited medication while enrolled in the study. (Appendix B: complete list of prohibited medications).

9. Non-English speakers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
nPEP Failure | 4 months active study participation
  HIV sero-conversion during study participation following high risk exposure that occured within 72 hours of study product initiation.
Safety and Tolerability assessed as Adverse Events and Safety Lab Evaluation | 4 months active study participation
  The following AEs will be evaluated: Diarrhea, Fatigue, Nausea/Vomiting, Headache, Dizziness, Body/Muscle/Joint pain

SECONDARY OUTCOMES:
Adherence and Acceptability assessed as study product completion rate | 4 months of active study participation or 28 days of study product use
  Completion of Study Product as Prescribed; Stopped or Modified Study Product, Lost to Follow Up

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H Mayer, MD, Principal Investigator — Fenway Health
Locations (1):
- Fenway Community Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mayer KH, Gelman M, Holmes J, Kraft J, Melbourne K, Mimiaga MJ. Safety and Tolerability of Once Daily Coformulated Bictegravir, Emtricitabine, and Tenofovir Alafenamide for Postexposure Prophylaxis After Sexual Exposure. J Acquir Immune Defic Syndr. 2022 May 1;90(1):27-32. doi: 10.1097/QAI.0000000000002912. PMID 34991141